CLINICAL TRIAL: NCT06245603
Title: A Study to Evaluate Efficacy and Safety of Hydeal Cyst® Intravesical Instillations in Patients Treated With Intravesical Chemotherapy or Immunotherapy in Non-muscle Invasive Bladder Cancer
Acronym: Hydeal Cyst
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Collaborators: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOV-NMIBC-01-2022-HydealCyst
Record Dates: First submitted 2024-01-19; First posted 2024-02-07 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-06

CONDITIONS: Non-muscle Invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Multicentre open-label, controlled, randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (interventional arm) (Experimental): patients receive Hydeal Cyst intravesical instillations during the BCG or MMC therapy period.
  Interventions: Device: Hydeal Cyst®
- Arm B (control arm) (No Intervention): patients receive only standard therapy (BCG or MMC).

INTERVENTIONS:
Device: Hydeal Cyst® — BCG or MMC will be started within 1-2 weeks from randomization (within 12-14 weeks after TURB).
  BCG or MMC will be administered once a week by intravesical instillation: BCG will be abministered for 6 weeks and MMC for 8 weeks. (induction cycles) Before instillations a physical examination will be performed and symptoms evaluated: changes from baseline and abnormalities will be recorded in patient notes.
  IPSS questionnaire and QoL questionaire will be administered to the patient at week 1, 4 and 6/8 (6 for BCG and 8 for MMC) of treatment.
  48 hours after post BCG or MMC intravesical instillation, patients of Arm A will undergo Hydeal Cyst intravesical instillation.
  BCG patiens will received 6 Hydeal Cyst intravesical instillation; MMC patiens will received 8 Hydeal Cyst intravesical instillation.
  Arms: Arm A (interventional arm)

SUMMARY:
Prior to performing any study specific procedure (including screening procedures to determine eligibility), a signed consent form will be obtained for each subject. Patients will be enrolled in the study only if they meet all the inclusion criteria and none of the exclusion criteria.

Prior to perform any study specific procedure (including screening procedures to determine eligibility), a signed informed consent form will be obtained for each subject. The informed consent form will describe the purpose of the study, the procedures to be followed, and the risk and benefits of participation. The investigator will conduct the informed consent discussion and will check that the subject comprehends the information provided and will answers any questions about the study. Consent will be voluntary and free from coercion. The investigator that will conduct the consent discussion will also sign the informed consent form. A copy of the informed consent form will be given to the subject and the fact that the subject has been consented to the study will be documented in the subject's record. When all the inclusion and exclusion criteria have been addressed and the eligibility of the subject confirmed, the subject may be enrolled in the study.

The following activities and/or assessments will be performed during screening, prior the treatment period start: demographic, medications related to the disease or symptoms and cancer history data collection; Urine-colture; randomization; Questionnaires QoL e IPSS.

BCG or MMC will be started within 1-2 weeks from randomization (within 12-14 weeks after TURB).

BCG or MMC will be administered once a week by intravesical instillation: BCG will be abministered for 6 weeks and MMC for 8 weeks. (induction cycles) Before instillations a physical examination will be performed and symptoms evaluated: changes from baseline and abnormalities will be recorded in patient notes.

IPSS questionnaire and QoL questionaire will be administered to the patient at week 1, 4 and 6/8 (6 for BCG and 8 for MMC) of treatment.

48 hours after post BCG or MMC intravesical instillation, patients of Arm A will undergo Hydeal Cyst intravesical instillation.

BCG patiens will received 6 Hydeal Cyst intravesical instillation; MMC patiens will received 8 Hydeal Cyst intravesical instillation.

After 2 weeks from BCG or MMC instillation end, IPSS e QoL questionaires will be administered and a control urino-colture will be executed.

After 6 and 18 weeks from instillation therapy end, a control visit will be made.

A physical examination will be performed and symptoms evaluated: changes from baseline and abnormalities will be recorded in patient notes.

Control cystoscopy and urino-colture will be executed (as for clinical practice) and IPSS and quality of life evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* ECOG PS 0-2
* Histologically confirmed diagnosis of non-muscle invasive bladder cancer, naïve and recurrent.
* Patients candidate to BCG or MMC intravesical induction therapy.
* Transurethral resection (TURB/re-TURB when indicated) performed in the last 12 weeks.
* IPSS score ≤19
* Negative urine culture within 2 weeks before T0
* For women who are not postmenopausal (i.e., < 1 year after last menstruation) or surgical-ly sterile (absence of ovaries and/or uterus) and who are sexually active: agreement to use an adequate method of contraception (oral contraceptives, intrauterine contraceptive de-vice, or barrier method of contraception in conjunction with spermicidal jelly) during the study period
* Signed the study informed consent prior to any study specific procedures.
* Will and ability to comply with the protocol

Exclusion Criteria:

* Upper urinary tract urothelial carcinoma (UTUC); bladder diverticula; urethral stenosis; difficult catheterization; reduced bladder compliance; increased bladder compliance; post-voiding residue > 150 ml;
* Surgery or invasive procedures planned during the study and interfering with evaluation about efficacy and safety of it.
* Female patients with child-bearing potential must not be pregnant or lactating, or not willing to use adequate contraception for the duration of study
* Pelvic radiotherapy within 24 weeks prior to the beginning of the study treatment.
* Urinary tract infection requiring antibiotics
* Have a known hypersensitivity to any substance present in the investigational device.
* Neurogenic bladder
* Any condition for that, in the opinion of the Investigator, participation would not be in the best interest of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Lower urinary tract symptoms | From the date of randomization up to 22 weeks
  Lower urinary tract symptoms will be evaluated by the IPSS questionnaire (score 0-35) at baseline and follow-up visits. Difference from baseline will be calculated at two weeks after the end of induction cycle of intravesical instillation.

SECONDARY OUTCOMES:
Recurrence free survival (RFS) | From the date of randomization up to 22 weeks
  The recurrence free survival (RFS) will be determined as the time from the date of randomization to the date of clinical disease recurrence. Patients without a RFS event at the time of analysis will be censored at the date of last assessment
Progression free survival (PFS) | From the date of randomization up to 22 weeks
  The progression free survival (PFS) will be determined as the time from the date of randomization to the date of clinical disease progression. Patients without a PFS event at the time of analysis will be censored at the date of last assessment
Toxicity during the treatment | From the date of randomization up to 22 weeks
  Toxicity during the treatment will be recorded and graded according to the NCI-Common Terminology Criteria for Adverse Events (CTCAE) v.5. Grade refers to the severity of the adverse event. A grading (severity) scale is provided for each adverse event term. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE.
Quality of Life assessment | From the date of randomization up to 22 weeks
  Quality of Life will be evaluated at randomization (T0), at weeks 4 and 6/8 (T6 for BCG/T8 for MMC) of instillation treatment and during follow-up period (weeks 2, 6 and 12 after instillation treatment end). QoL will be assessed throught the FACT-Bl questionnaire.

CONTACTS AND LOCATIONS:
Locations (9):
- Italy (9):
  - Humanitas Gavezzeni-Bergamo, Bergamo
  - Ospedale Sant'Orsola - Malpighi, Bologna
  - Policlinico Ospedali Riuniti - Foggia, Foggia
  - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda Ospedale Università Padova, Padua
  - Ospedali Riuniti Padova Sud, Padua
  - Policlinico Paolo Giaccone, Palermo
  - Ospedale Santa Maria della Misericordia - ASU FC, Udine
  - Azienda Ospedaliera Universitaria Integrata - Verona, Verona

IPD SHARING:
Plan to Share IPD: No